CLINICAL TRIAL: NCT04710069
Title: Randomized Controlled Trial for Postoperative opt-in Narcotic Treatment in Outpatient Endocrine Surgery
Brief Title: Postoperative Opt-In Narcotic Treatment Study
Acronym: POINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, James Wu, MD, Dr. James Wu, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-001702
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain; Narcotic Use; Analgesia; Endocrine Surgery; Opioid Use; Opioid Abuse
Keywords: Postoperative Pain; Narcotic Use; endocrine surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Attending surgeons are not aware of participant treatment arm until after the participant undergoes their operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control/Usual Care (No Intervention): standard treatment of postoperative pain, which involves automatic prescription of a narcotic pain medication regimen after surgery,
- Opt-in/POINT (Experimental): An opt-in program (POINT), which requires the patient to consent to receiving a prescription for narcotics
  Interventions: Behavioral: POINT

INTERVENTIONS:
Behavioral: POINT — Patients randomized to the POINT program will be given preoperative counseling on adverse effects of opioids and expectations will be set that most patients do not require opioids for pain control after endocrine surgery, they will receive the info in writing afterwards as well. These patients will also be shown a short instructional video reiterating the counseling provided in the preoperative clinic visit. Information in the video will pertain to the expected pain after surgery, the over-the-counter options for pain control, the risks and side effects of using opioids, and reassurances that opioids may be prescribed at any time after discharge if pain is unmanageable. After the video, the patient will be provided with paperwork, requiring patient consent/signature to receive opioids if they opt into narcotic treatment. They will not be provided with a narcotic prescription if consent is not explicitly provided.
  Other Names: Opt-in
  Arms: Opt-in/POINT

SUMMARY:
pills go unused, generating waste and leaving an opportunity for misuse and abuse.

In a recent study, researchers let patients choose what medications to go home with after surgery. After their thyroid or parathyroid surgery, 96% of patients declined narcotic pain medication. They preferred to manage their pain with acetaminophen instead. Giving patients counseling and empowering them to choose significantly reduces the amount of opioids prescribed and wasted.

The aim of our study is to compare a similar "opt-in" protocol for narcotics to usual care (where patients are routinely discharged with opioids). We would elaborate upon the aforementioned study by studying patient pain scores on a more granular level once they return home.

Our study will be designed as a randomized, controlled trial. When adult patients consent for a thyroid or parathyroid surgery, they will be asked to participate in the study. Patients who are currently using narcotics would be excluded. We would then randomize participants to the "opt-in" protocol versus being provided with a standard opioid prescription after surgery. Patients in the opt-in protocol will be recommended a pain treatment regimen with over-the-counter medications, such as acetaminophen or ibuprofen. These patients will be reassured that if their pain is uncontrolled after discharge, a narcotic prescription will be called in to their pharmacy if requested.

We will assess patient pain scores and medication use in the recovery area using the electronic medical record. We will collect data on patient pain scores and medication use after discharge on a daily basis via phone call or electronically transmitted survey. We will also evaluate patients at the time of their follow-up visits. Any patient phone calls will be routed to study personnel who will fill narcotic prescription requests if requested. Finally, among patients who do receive an opioid prescription, we will track their opioid consumption.

DETAILED DESCRIPTION:
Due to the current opioid epidemic, there has been increased focus on the prescribing patterns of physicians and greater incentive to reduce the amount of narcotic pain medication prescribed.

A prospective study was recently published in Annals of Surgery by Ruffolo et al. which described an opt-in narcotic treatment program for 216 patients who underwent outpatient endocrine cervical surgery (1). Patients were counseled in the pre-operative visit that after the surgery, they would be provided the option of narcotic pain medication versus over-the-counter medication. Prior to discharge, patients were evaluated by a member of the surgical team and offered a choice of postoperative pain medications. The study found only 4% of patients requested narcotic pain medication and achieved a 96.6% reduction in postoperative narcotic use. No patients called in to request narcotic pain medication after discharge.

The study participants were compared to a retrospective cohort of patients who were given narcotic medication postoperatively as the default option. There have been no randomized controlled trials comparing the two pain medication strategies in outpatient cervical endocrine surgery. Additionally, in that study, the level of postoperative pain was not fully assessed and quality of life measures were not studied.

In our institutional practice, having a member of the surgical team visit the patient at the bedside to assess pain level is not part of the standard postoperative work flow, given that the operative team is usually operating at the time the patient is discharged. In order to assess the feasibility of implementing such a program within our practice, we plan to develop alternative methods of presenting the decision for postoperative pain treatment in the immediate postoperative period that fits into our standard practice.

Significance:

Given the current health care and political climate, there has been increasing focus on reducing the amount of narcotics prescribed by health care providers. Based on the results of the above cited study, we believe implementing an opt-in program at UCLA will also significantly decrease the amount of opioids prescribed for postoperative pain. However, we will improve upon that study but assessing pain levels in the week immediately after surgery to ensure patients are not suffering from excessive pain levels at home without notifying providers, and compare these pain levels to patients who are randomized to standard postoperative care (automatically dispensed with a narcotic prescription). We will also assess quality of life measures after surgery to compare the impact of pain management strategy on the postoperative experience.

Ruffolo et al. demonstrated the feasibility in reducing the amount of narcotics prescribed by a significant level by initiating an opt-in program and empowering patients to make their own health care decisions. Incorporating this type of program into the standard operative work flow will maintain efficiency while working towards the goal of reducing narcotic usage. If we can demonstrate the feasibility of implementing such an opt-in program within the section of Endocrine Surgery, expanding the program to other divisions of ambulatory surgery in different surgical subspecialties may also be possible.

1. Ruffolo LI, Jackson KM, Juviler P, et al. Narcotic Free Cervical Endocrine Surgery: A Shift in Paradigm. Ann Surg. 9000;Publish Ahead of Print.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for outpatient parathyroidectomy, thyroidectomy or neck dissection Patients aged 18 or older English-speaking: Our provided materials (video instruction, written instructions, survey material) will be in English and we want to ensure clear communication with our study subjects. Once we have demonstrated feasibility of such an opt-in policy with our English-speaking subjects, we will expand our materials to additional languages.

Exclusion Criteria:

* Prior history of narcotic use Inpatient admission after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | Postoperative Day 0-7
  Pain scores will be compared using regression analysis and t-tests.
oral morphine equivalents consumed | Postoperative Day 0-7
  Possible predictors for narcotic use or higher pain scores will be assessed, including age, sex, type of surgery and preoperative questionnaire (PHQ-9) score using a mixed-effects model.

SECONDARY OUTCOMES:
Postoperative Day 0-7 | Postoperative Day 7
  Possible predictors for narcotic use or higher pain scores will be assessed, including age, sex, type of surgery and preoperative questionnaire (PHQ-9) score using a mixed-effects model.

CONTACTS AND LOCATIONS:
Overall Officials: James Wu, MD, Principal Investigator — University of California, Los Angeles; Michael W Yeh, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruffolo LI, Jackson KM, Juviler P, Kaur R, Chennell T, Glover DM, Linehan DC, Moalem J. Narcotic Free Cervical Endocrine Surgery: A Shift in Paradigm. Ann Surg. 2021 Aug 1;274(2):e143-e149. doi: 10.1097/SLA.0000000000003443. PMID 31356280
- [Derived] Zhu CY, Schumm MA, Hu TX, Nguyen DT, Kim J, Tseng CH, Lin AY, Yeh MW, Livhits MJ, Wu JX. Patient-Centered Decision-making for Postoperative Narcotic-Free Endocrine Surgery: A Randomized Clinical Trial. JAMA Surg. 2021 Nov 1;156(11):e214287. doi: 10.1001/jamasurg.2021.4287. Epub 2021 Nov 10. PMID 34495283